CLINICAL TRIAL: NCT01893229
Title: Comparative Efficacy and Acceptability of Lithium, Valproate, Oxcarbazepine, Quetiapine, Olanzapine, and Ziprasidone in Bipolar I Disorder, Manic or Mixed Phase
Brief Title: Comparative Efficacy and Acceptability of Antimanic Drugs in Acute Mania
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guiyun Xu (Other Government)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Sponsor-Investigator, Guiyun Xu, Associate Professor, Guangzhou Psychiatric Hospital
Organization: Guangzhou Psychiatric Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20120509
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Comparative Effectiveness Research; Therapeutics; Patient Dropouts
MeSH Terms: conditions — Bipolar Disorder; Patient Dropouts | interventions — Lithium; Lithium Carbonate; Valproic Acid; Oxcarbazepine; Quetiapine Fumarate; Olanzapine; ziprasidone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Valproate (Experimental): Name: Valproate; dosage form: tablet, 250mg; dosage and frequency: 800mg-- 1200mg/d; duration: 6 weeks.
  Interventions: Drug: Valproate
- Oxcarbazepine (Experimental): Name: Oxcarbazepine, dosage form: 300mg, tablet; dosage and frequency: 600-1200mg/d; duration: 6 weeks
  Interventions: Drug: Oxcarbazepine
- Quetiapine (Experimental): name: Quetiapine, dosage form: 200mg,tablet; dosage and frequency: 600mg-- 800mg/d; duration: 6 weeks
  Interventions: Drug: Quetiapine
- Olanzapine (Experimental): Name: Olanzapine, dosage form: 5mg tablet; dosage and frequency: 10mg--20mg/d; duration: 6 weeks
  Interventions: Drug: Olanzapine
- Ziprasidone (Experimental): Name: Ziprasidone, dosage form: 10mg tablet; dosage and frequency: 80mg-160mmg/d; duration: 6 weeks
  Interventions: Drug: Ziprasidone
- Lithium (Experimental): name: lithium; dosage form: 250mg Tablet; dosage and frequency: 750mg-2000mg/d;serum Li level: 0.6mmol-1.2mmol/L; duration: 6 weeks
  Interventions: Drug: Lithium

INTERVENTIONS:
Drug: Lithium — Lithium is used as a mood stabiliser
  Other Names: lithium Carbonate
  Arms: Lithium
Drug: Valproate — Valproate is used as a mood stabiliser
  Other Names: Depakote
  Arms: Valproate
Drug: Oxcarbazepine — Oxcarbazepine is used as a mood stabiliser
  Other Names: Trileptal
  Arms: Oxcarbazepine
Drug: Quetiapine — Quetiapine is used as a mood stabiliser
  Other Names: SEROquel
  Arms: Quetiapine
Drug: Olanzapine — Olanzapine is used as a mood stabiliser.
  Other Names: Zyprexa；
  Arms: Olanzapine
Drug: Ziprasidone — Ziprasidone is used as a mood stabiliser
  Other Names: Geodon
  Arms: Ziprasidone

SUMMARY:
Background:

Bipolar disorder is one of the most common mental illnesses affecting 1%-4% of the population, and one of the leading causes of worldwide disability. Mania is a condition of excessively elevated mood, characterizes bipolar disorder, and usually is a main cause of hospitalization. Mood stabilisers and antipsychotic drugs have long been the maintenance treatment of acute mania with and without psychotic symptoms. Though clinical trails have been demonstrated that these drugs are individually more effective than placebo in the relatively long term (e.g 4, 8 weeks). However, in the pragmatic practice, patient at acute mania urgently want to see the effectiveness, and psychiatrist under great pressure and are in great need to evaluate the very short-term effectiveness (e.g one week). If the first attempted antimanic drug fails, psychiatrist need the evidence that which medication should be to added on or switch to.

Objectives:

one main aim is to rank the short-term ( e.g.one and two week) effectiveness and acceptability of the common anti-mania drugs, including Lithium, Valproate, Oxcarbazepine, Quetiapine, Olanzapine, or Ziprasidone. Secondary aim is to investigate which medication to add on for non-responders or switch to.

Methods:

The study setting: it is expected that 120 subjects with a diagnose of DSM-IV bipolar I disorder will be recruited from Guangzhou Psychiatric Hospital, the earliest psychiatric hospital in the history of China established by Dr.J. G. Kerr in 1898.

Design:This study is a randomized, controlled trial. Participants with a Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis of bipolar I disorder, manic or mixed episode will be randomly assigned to a treatment of Lithium, Valproate, Oxcarbazepine, Quetiapine, Olanzapine, or Ziprasidone. In the following conditions, participants will take another antimanic drug as a combination medication: 1) those who have a reduction in YMRS scores less than 25% after one week of treatment; 2) those who have a reduction in YMRS scores less than 50% after two weeks of treatment; or 3) those who have a increase in YMRS more than 30% at day 4. An antipsychotic (Quetiapine, Olanzapine, and Ziprasidone) will be added on for those who use lithium, Valproate or Oxcarbazepine as a first attempted medication; while Lithium, Valproate, or Oxcarbazepine will be added on for those who use an antipsychotic as a first attempted medication. Those participants who are recognized as non-response/partial response to two combined medications after 6 weeks of treatment will switch to Modified Electroconvulsive Therapy (MECT).

Measures: Primary outcome measures are change scores on the Young Mania Rating Scale (YMRS) and dropout rates. Secondary outcome measures include Clinical Global Impressions (CGI) Scale, Global Assessment Scale (GAS), Treatment Emergent Symptom Scale (TESS), and Brief Psychiatric Rating Scale (BPRS).

Response criteria: <25% reduction in YMRS scores or >=4 scores of CGI is defined as non-response. 25-49% reduction in YMRS scores from baseline as well as <=3 scores of Clinical General Impression (CGI) is recognized as partial response.>= 50% reduction in YMRS as well as 1 (very much improved) or 2 scores (much improved) of CGI is recognized as response. Remission is defined as a YMRS score <=12 and CGI score equal to 1 or 2.

DETAILED DESCRIPTION:
Background:

Bipolar disorder is one of the most common mental illnesses affecting 1%-4% of the population, and one of the leading causes of worldwide disability. Mania is a condition of excessively elevated mood, characterizes bipolar disorder, and usually is a main cause of hospitalization. Mood stabilisers and antipsychotic drugs have long been the maintenance treatment of acute mania with and without psychotic symptoms. Though clinical trails have been demonstrated that these drugs are individually more effective than placebo.However, in the pragmatic practice, patient at acute mania urgently want to see the effectiveness, and psychiatrist under great pressure and are in great need to evaluate the very short-term effectiveness (e.g one week). If the first attempted antimanic drug fails, psychiatrist need the evidence that which medication should be to added on or switch to.

Objectives:

one main aim is to rank the short-term ( e.g.one and two week) effectiveness and acceptability of the common anti-mania drugs, including Lithium, Valproate, Oxcarbazepine, Quetiapine, Olanzapine, or Ziprasidone. Secondary aim is to investigate which medication to add on for non-responders or switch to.

Methods:

The study setting: it is expected that 120 subjects with a diagnose of DSM-IV bipolar disorder will be recruited from Guangzhou Psychiatric Hospital, the earliest psychiatric hospital in the history of China established by Dr.J. G. Kerr in 1898.

Design:This study is a randomized, controlled trial, consisting two phase. 120 participants with a Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis of bipolar I disorder, manic or mixed phase will be randomly assigned to a treatment of Lithium, Valproate, Oxcarbazepine, Quetiapine, Olanzapine, or Ziprasidone. The period from starting dose to effective dose for each drug is within 2 days, and the effective doses for these drugs are described as follow: Lithium, 750mg-2000mg/d, serum Li level: 0.6mmol-1.2mmol/L; Valproate, 800mg-- 1200mg/d, serum Valproate level: 70-120ug/ml; Oxcarbazepine, 600-1200mg/d; Quetiapine, 600mg--800mg/d; Olanzapine, 10mg-- 20mg/d; Ziprasidone, 80mg-160mmg/d.

In the following conditions, participants will take a another antimanic drug as a combination medication: 1) those who have a reduction in YMRS scores less than 25% after one week of treatment; 2) those who have a reduction in YMRS scores less than 50% after two weeks of treatment; or 3) those who have a increase in YMRS more than 30% at day 4. An antipsychotic (Quetiapine, Olanzapine, and Ziprasidone) will be added on for those who use lithium, Valproate or Oxcarbazepine as a first attempted medication; while Lithium, Valproate, or Oxcarbazepine will be added on for those who use an antipsychotic as a first attempted medication. Those participants who are recognized as non-response/partial response to two combined medications after 6 weeks of treatment will switch to Modified Electroconvulsive Therapy (MECT).

Measures: Primary outcome measures are change scores on the Young Mania Rating Scale (YMRS) and dropout rates. Secondary outcome measures include Clinical Global Impressions (CGI) Scale, Global Assessment Scale (GAS), Treatment Emergent Symptom Scale (TESS), and Brief Psychiatric Rating Scale (BPRS).

Response criteria: <25% reduction in YMRS scores or >=4 scores of CGI is defined as non-response. 25-49% reduction in YMRS scores from baseline as well as <=3 scores of Clinical General Impression (CGI) is recognized as partial response.>= 50% reduction in YMRS as well as 1 (very much improved) or 2 scores (much improved) of CGI is recognized as response. Remission is defined as a YMRS score <=12 and CGI score equal to 1 or 2.

ELIGIBILITY:
Inclusion Criteria:

* with a diagnosis of bipolar I disorder, manic or mixed phase
* equal or more than 18 scores in Young Mania Rating Scale (YMRS)

Exclusion Criteria:

* Serious general medical illness
* pregnancy and lactation
* given long-acting antipsychotic drug within the last two month
* endocrine disease( e.g.Diabetes and thyrotoxicosis)
* given thyroxine therapy within the last three months or is being given hormone therapy
* sexually active and not using contraceptives

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Young Mania Rating Scale at 2 weeks and 6 weeks | Baseline, 2 weeks and 6 weeks
  Young Mania Rating Scale is used to assess hypomania/mania symptoms
rate of dropout (treatment discontinuation) | 1,2,4,6 weeks
  to compare the rates of treatment discontinuation of different drugs because of side effect or effectiveness

SECONDARY OUTCOMES:
Clinical Global Impressions (CGI) Scale | baseline, 2 weeks, 4 weeks, and 6 weeks
  Clinical Global Impressions (CGI) Scale is used to assess the patient's global functioning prior to and after initiating a study medication. The CGI provides an overall clinician-determined summary measure, taking into account all available information, including a knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function
Brief Psychiatric Rating Scale | baseline, 2, 3, 4 and 6 weeks
  Brief Psychiatric Rating Scale is used to assess psychotic symptoms.
Global Assessment Scale | baseline, 2, 3, 4 and 6 weeks
  Global Assessment Scale is a numeric scale (1 through 100) used by mental health clinicians to rate the general functioning.
Treatment Emergent Symptom Scale | 2, 3, 4 and 6 weeks
  Treatment Emergent Symptom Scale is used to assess the adverse event of the drug.
Hamilton Anxiety Rating Scale | baseline, 2, 3, 4, and 6 weeks
  Hamilton Anxiety Rating Scale is used to assess anxious symptoms
Hamilton Depression Rating Scale | baseline, 2, 3, 4, and 6 weeks
  Hamilton Depression Rating Scale is used to assess the depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Guinyun Xu, M.D, Principal Investigator — Guangzhou Psychiatric Hospital; Kangguang Lin, M.D, Principal Investigator — The University of Hong Kong
Locations (1):
- Guangzhou Psychiatric Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Murray CJ, Lopez AD. Global mortality, disability, and the contribution of risk factors: Global Burden of Disease Study. Lancet. 1997 May 17;349(9063):1436-42. doi: 10.1016/S0140-6736(96)07495-8. PMID 9164317
- [Background] Tarr GP, Glue P, Herbison P. Comparative efficacy and acceptability of mood stabilizer and second generation antipsychotic monotherapy for acute mania--a systematic review and meta-analysis. J Affect Disord. 2011 Nov;134(1-3):14-9. doi: 10.1016/j.jad.2010.11.009. Epub 2010 Dec 9. PMID 21145595
- [Background] Correll CU, Sheridan EM, DelBello MP. Antipsychotic and mood stabilizer efficacy and tolerability in pediatric and adult patients with bipolar I mania: a comparative analysis of acute, randomized, placebo-controlled trials. Bipolar Disord. 2010 Mar;12(2):116-41. doi: 10.1111/j.1399-5618.2010.00798.x. PMID 20402706
- [Background] Cipriani A, Barbui C, Salanti G, Rendell J, Brown R, Stockton S, Purgato M, Spineli LM, Goodwin GM, Geddes JR. Comparative efficacy and acceptability of antimanic drugs in acute mania: a multiple-treatments meta-analysis. Lancet. 2011 Oct 8;378(9799):1306-15. doi: 10.1016/S0140-6736(11)60873-8. Epub 2011 Aug 16. PMID 21851976
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders. 4th ed. text revision. Washington (DC): American Psychiatric Association; 2000.
- [Background] Zhang L, Ning Y. Guangzhou psychiatric hospital: the oldest psychiatric hospital in china. Psychiatry (Edgmont). 2010 Jun;7(6):53-4. PMID 20622947